CLINICAL TRIAL: NCT02352376
Title: Effects of Non Invasive Ventilation on Heart Rate Variability After Coronary Bypass Grafting: Comparison Between Different Ventilator
Brief Title: Noninvasive Ventilation After Coronary Bypass Grafting
Acronym: Physiotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Célia Regina Lopes, EFFECTS OF NON INVASIVE VENTILATION ON HEART RATE VARIABILITY AFTER CORONARY BYPASS GRAFTING: COMPARISON BETWEEN DIFFERENT VENTILATORS, Federal University of Uberlandia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11104413.6.0000.5152
Record Dates: First submitted 2014-11-10; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Coronary Artery Bypass
Keywords: Noninvasive ventilation; Heart rate variability; Thoracic surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional ventilator (Other): 30 minutes of non-invasive ventilation was performed with conventional ventilator.The order of the procedures was determined by randomization.
  Interventions: Other: Conventional ventilator; Other: Specific ventilator
- Specific ventilator (Other): 30 minutes of non-invasive ventilation was performed with specific respirator. The order of the procedures was determined by randomization.
  Interventions: Other: Conventional ventilator; Other: Specific ventilator

INTERVENTIONS:
Other: Conventional ventilator — A ventilator designed for invasive ventilation was used has mode non-invasive ventilation with leakage compensation (50% of the predetermined tidal volume).
Other: Specific ventilator — A ventilator was used designed for non-invasive ventilation has an algorithm that calculates the loss of pressure and automatically compensates for leak

SUMMARY:
This is a prospective, quantitative, randomized, crossover study. Were included in this study 10 people in the Intensive Care Unit at University Hospital in Uberlandia, on the first day of the postoperative coronary artery bypass graft (CABG). For data collection was performed randomization on the block (2: 4), to determine the first technique to be used and then a wash-out period of one hour was allowed for the research subject reaches the systemic arterial pressure, heart rate, respiratory rate and oxygen saturation baseline. And after, for cross-over, the second technique was performed. Non-invasive ventilation was performed for 30 minutes each ventilator. All subjects underwent noninvasive ventilation using two models of ventilators, they are conventional (designed for invasive ventilation but is also used in non-invasive ventilation mode) and specific (designed for non-invasive ventilation). Hemodynamic, autonomic and respiratory variables are monitored. We use the hypothesis that non-invasive ventilation performed with two fan models can alter autonomic function and that there is hemodynamic changes related to autonomic function in different ventilators in postoperative coronary artery bypass grafting.

DETAILED DESCRIPTION:
Background: The patients in postoperative coronary artery bypass graft (CABG) have impaired cardiac autonomic function. However, no studies have evaluated the influence of different ventilators during noninvasive ventilation (NIV) in the autonomic modulation associated with hemodynamic changes. Objective: Evaluate the autonomic behavior and hemodynamic changes during the execution of the NIV with two models of mechanical ventilators in subjects after CABG. Material and Methods: This is quantitative randomized, prospective, crossover study. The subjects were selected on first day postoperatively CABG and was performance NIV procedure using two different ventilators: conventional ventilator and specific ventilator for the use of NIV for 30 minutes, each. Block randomization was used to determine the technique that begins to approach then by crossover, perform the sequential technique. The heart rate variability (HRV), heart rate, respiratory rate, oxygen peripheral saturation and arterial pressure were evaluated before procedure, in the instants 5, 10, 15, 20, 25, 30 minutes during NIV each and 15 minutes after the end of the NIV application. HRV was evaluated using the time and frequency domain.

ELIGIBILITY:
Inclusion criteria

* Age over 18 years .Who were breathing spontaneously with peripheral oxygen saturation (SpO2) ≥ 90% and supplemental oxygen ≤ 3 l / min.
* Indication for use of NIV

Exclusion criteria

* Hemodynamic instability with hypertensive response being considered systolic blood pressure (SBP) greater than 180 mmHg and diastolic blood pressure (DBP) greater than 110 mmHg, or difference in SBP and DBP less than 20 mmHg or framework shock considering SBP <90 mmHg and / or DBP <50 mmHg, since the normal SBP were between 90-130 mmHg and DBP 60-90 mmHg
* Presence of active cardiac pacemaker
* Invasive mechanical ventilation more than 24 hours
* Use of intra aortic balloon
* Postoperatively Myocardial infarction after surgery
* Ineffective cough with bronchial hypersecretion
* Inability to adequately swallowing and/or protect the airway
* Abdominal distension
* Nausea
* Vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Variability of heart rate front the use of noninvasive ventilation in two different ventilators in patients after cardiac surgery, measured by Polar RS800 CX. | 3 hours
  The autonomic variables evaluated are: standard deviation of all normal RR intervals recorded in a time interval (SDNN); standard deviation of the mean of normal RR intervals every 5 minutes at a time, expressed in milliseconds (SDANN); percentage of R-Ri with adjacent difference of duration greater than 50 milliseconds (pNN50) and the square root of the average squared difference between the adjacent R-Ri normal in a period of time, expressed in milliseconds (rMSSD). All variables will be assessed by Polar RS800CX

SECONDARY OUTCOMES:
Change in the indices of variability of heart rate, systolic blood pressure, diastolic blood pressure and heart rate during noninvasive ventilation with two models of ventilatotors in patients after cardiac surgery. | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Valdeci C Dionísio, Dr., Principal Investigator — Federal University of Uberlandia

REFERENCES:
- [Result] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Result] Carnevali L, Sgoifo A. Vagal modulation of resting heart rate in rats: the role of stress, psychosocial factors, and physical exercise. Front Physiol. 2014 Mar 24;5:118. doi: 10.3389/fphys.2014.00118. eCollection 2014. PMID 24715877
- [Result] Pantoni CB, Di Thommazo L, Mendes RG, Catai AM, Luzzi S, Amaral Neto O, Borghi-Silva A. Effects of different levels of positive airway pressure on breathing pattern and heart rate variability after coronary artery bypass grafting surgery. Braz J Med Biol Res. 2011 Jan;44(1):38-45. doi: 10.1590/s0100-879x2010007500129. Epub 2010 Nov 19. PMID 21085891
- [Result] Ozyilmaz E, Ugurlu AO, Nava S. Timing of noninvasive ventilation failure: causes, risk factors, and potential remedies. BMC Pulm Med. 2014 Feb 13;14:19. doi: 10.1186/1471-2466-14-19. PMID 24520952
- [Result] Sasaki K, Maruyama R. Consciously controlled breathing decreases the high-frequency component of heart rate variability by inhibiting cardiac parasympathetic nerve activity. Tohoku J Exp Med. 2014 Jul;233(3):155-63. doi: 10.1620/tjem.233.155. PMID 24965685
- [Result] Radaelli A, Raco R, Perfetti P, Viola A, Azzellino A, Signorini MG, Ferrari AU. Effects of slow, controlled breathing on baroreceptor control of heart rate and blood pressure in healthy men. J Hypertens. 2004 Jul;22(7):1361-70. doi: 10.1097/01.hjh.0000125446.28861.51. PMID 15201553
- [Result] Pinsky MR. Cardiovascular issues in respiratory care. Chest. 2005 Nov;128(5 Suppl 2):592S-597S. doi: 10.1378/chest.128.5_suppl_2.592S. PMID 16306058
- [Result] Zhu GF, Wang DJ, Liu S, Jia M, Jia SJ. Efficacy and safety of noninvasive positive pressure ventilation in the treatment of acute respiratory failure after cardiac surgery. Chin Med J (Engl). 2013 Dec;126(23):4463-9. PMID 24286408
- [Result] Zarbock A, Mueller E, Netzer S, Gabriel A, Feindt P, Kindgen-Milles D. Prophylactic nasal continuous positive airway pressure following cardiac surgery protects from postoperative pulmonary complications: a prospective, randomized, controlled trial in 500 patients. Chest. 2009 May;135(5):1252-1259. doi: 10.1378/chest.08-1602. Epub 2008 Nov 18. PMID 19017864
- [Result] Yang LX, Zhou YJ, Wang ZJ, Li YP, Chai M. Impact of invasive treatment strategy on health-related quality of life six months after non-ST-elevation acute coronary syndrome. J Geriatr Cardiol. 2014 Sep;11(3):206-11. doi: 10.11909/j.issn.1671-5411.2014.03.003. PMID 25278968
- [Result] Yan TD, Padang R, Poh C, Cao C, Wilson MK, Bannon PG, Vallely MP. Drug-eluting stents versus coronary artery bypass grafting for the treatment of coronary artery disease: a meta-analysis of randomized and nonrandomized studies. J Thorac Cardiovasc Surg. 2011 May;141(5):1134-44. doi: 10.1016/j.jtcvs.2010.07.001. Epub 2010 Dec 17. PMID 21167508